CLINICAL TRIAL: NCT05182320
Title: Multicenter, Prospective, Randomized, Comparative Study Measuring the Effects on Clinical Outcomes, Patient Satisfaction, Costs and Benefits of Combined Pre-, Intra- and Postoperative Patient Data for THA and TKA Patients Using an APP Based Sensor for Exercise Performance Before and After Operation
Brief Title: Study Measuring the Effects of Patient Data for Total Hip and Total Knee Arthroplasty Patients Using an APP Based Sensor for Home Exercise Performance Before and After Operation
Acronym: ORTHOPATH
Status: Withdrawn | Type: Observational
Why Stopped: contracts were not closed in time
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2108
Record Dates: First submitted 2021-12-01; First posted 2022-01-10 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee; Clinical Outcome; Patient Satisfaction; Treatment Cost
Keywords: randomized comparative study; clinical outcome; App based sensor; Home Exercise
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OrthoPath
  Interventions: Device: OrthoPath
- Control
  Interventions: Device: Control

INTERVENTIONS:
Device: OrthoPath — unilateral TKA and THA patients using the BPMpathway rehabilitation sensor system
  Groups: OrthoPath
Device: Control — unilateral TKA and THA patients not using the BPMpathway rehabilitation sensor system
  Groups: Control

SUMMARY:
Multicenter, Prospective, Randomized, Comparative Study Measuring the Effects on Clinical Outcomes, Patient Satisfaction, Costs and Benefits of Combined Pre-, Intra- and Postoperative Patient Data for THA and TKA Patients Using an APP Based Sensor for Home Exercise Performance Before and After Operation

ELIGIBILITY:
Inclusion Criteria:

* Primary, unilateral total knee and hip replacement patients
* Participant is min. 18 years of age
* Participant is able and willing to provide written informed consent
* Participant with ability to work with smart devices
* Participant having its own device (Apple iPhone or iPad with latest iOS version or Android tablet or smart phone min. Android version 6) and are able to handle the app and/or sensor

Exclusion Criteria:

* Pregnancy
* Participant has mental in capabilities - unable to give informed consent
* Participants who are unwilling or mentally and/or physically unable to adhere to study procedures
* Participant is having orthopaedic co-morbidities such as: previous HTO at indexed joint or prior UKA
* Flexion contracture > 15°
* Varus/valgus deformity > 10°
* Participant is having dementia or other cognitive impairment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary unilateral Total Knee and Hip Arthroplasty
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Osteoarthritis Outcome Score | 12 weeks after surgery
  The Patient self-assessed Injury and Osteoarthritis Outcome Scores for Knee (KOOS) and hip (HOOS) are joint-specific instruments:
  The KOOS evaluates both short-term and long-term consequences of knee injury. It holds 42 items in 5 separately scored subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL).
  The HOOS evaluates both short-term and long-term consequences of hip injury. It holds 5 separate patient-relevant dimensions: Pain (P), Symptoms (S), Activity limitations daily living (ADL), Function in sport and recreation (SP) and hip related quality of life (QOL).
  Both scores are percentage scores from 0 to 100, 0 representing extreme problems and 100 representing no problems.

SECONDARY OUTCOMES:
Patient satisfaction | 12 weeks after surgery
  Based on a single question patients are asked to grade their level of satisfaction with the methodology and rehabilitation procedure. Patients can choose between "very dissatisfied", "dissatisfied", "satisfied" or "very satisfied". The grades may be summarized as "satisfied" vs. "dissatisfied".
Patient User Experience | at final follow-up approx. 7 months after surgery
  A measurement just for the patients of the study group. The user feedback is collected at the endpoint
Patient compliance | at final follow-up approx. 7 months after surgery
  A measurement just for the patients of the study group. Data collection (Counting) how often patients use BPMpathway before and after operation to determine compliance with specification of using BPMpathway three times per day every day through data analytics
Economical [time and costs] | 12 weeks after surgery
  Comparing conventional rehabilitation methods and tele-rehabilitation under cost aspects enlarged by quality aspects such as acceptance and satisfaction degree of the patient
Course of Active Range of Motion | repeatedly from pre-op consultation until final follow-up approx. 7 months after surgery
  Study Group: Measured with BPMpathway sensor and app 3 times per day for the entire duration and measures with manual goniometer during all clinical visits (in 5° steps) Control Group: Measured with manual goniometer during all clinical visits (in 5°steps)
Development of Pain | repeatedly through study completion, an average of 7 months postoperatively.
  Study Group: Pain measured within BPMpathway app 3 times per day for the entire duration by Wong Baker Pain Score until post-operative follow-up meeting and during all clinical visits Control Group: Pain measured with Wong Baker Pain Scale during all clinical visits
  The Wong-Baker proves to be an inexpensive, yet easy to use, pain scale. The scale consists of six faces that range from no pain at all to the worst pain imaginable. The emotional faces range from smiling to grimacing.
Fatigue | at pre-operative consultation, post-operative consultation (12 weeks) and 6 months after surgery
  Study Group and Control Group: Measures with Fatigue Severity Scale. The Fatigue Severity Scale is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. It was originally devised for people with Multiple Sclerosis or systemic lupus erythematosus.
  The items are scored on a 7-point scale with 1=strongly disagree and 7=strongly agree; the minimum score is 9 and the maximum score is 63. The higher the score the greater the fatigue severity.
Radiographic Analysis | through study completion, an average of 7 months postoperatively
  Unless limited by patient or equipment constraints, all follow-up imaging exams will be obtained. Imaging will be used to evaluate the implant status as well as device condition and potential presence of device-related Adverse Events including fracture, wear, loosening or radiolucencies. X-rays are taken according to the radiographic protocol of the hospital and the set routine
Number of (Serious) Adverse Events | through study completion, an average of 7 months postoperatively
  During the course of the study, any upcoming intra- or postoperative (serious) adverse device events or effects related or not related to the product under investigation, will be documented in the dedicated Case Report Forms. The total number of AEs will be summarized and further evaluated by the sponsor and reported according to local legislation and necessity. Recorded complications will be categorized and analyzed in order to assess the safety of the investigational product

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Sportklinik Ravensburg GmbH & Co. KG, Ravensburg, Baden-Wurttemberg
  - RHÖN-KLINIKUM Campus Bad Neustadt, Bad Neustadt an der Saale

IPD SHARING:
Plan to Share IPD: No